CLINICAL TRIAL: NCT07026695
Title: Transcutaneous Electrical Vagus Nerve Stimulation for Suppression of Ventricular Arrhythmias
Brief Title: Transcutaneous Vagus Nerve Stimulation for Ventricular Arrhythmias
Acronym: TREAT-VT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 177627
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Premature Ventricular Complexes; Ventricular Tachycardia (VT); Ventricular Arrhythmias
Keywords: double-blinded; randomized; sham-controlled; crossover; prospective
MeSH Terms: conditions — Ventricular Premature Complexes; Tachycardia, Ventricular

STUDY DESIGN:
Intervention Model Description: Double-blinded, randomised, sham-controlled, crossover trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Phase (Active Comparator)
  Interventions: Device: transcutaenous vagal nerve stimulation
- Sham Phase (Sham Comparator)
  Interventions: Device: Sham transcutaenous vagal nerve stimulation

INTERVENTIONS:
Device: transcutaenous vagal nerve stimulation — Low level Stimulation of the Auricular Branch of the Vagal Nerve at the tragus
  Arms: Active Phase
Device: Sham transcutaenous vagal nerve stimulation — Sham treatment
  Arms: Sham Phase

SUMMARY:
Ventricular arrhythmias are abnormal heart rhythms that arise from the bottom chambers of the heart. They can cause debilitating symptoms when they occur intermittently (these are called premature ventricular ectopics or PVCs) and can be life-threatening when they occur continuously (called ventricular tachycardia or VT). These are the most common causes of sudden cardiac death, especially in patients with pre-existing heart disease.

They can be a result of overactivation of the sympathetic nervous system, and in extreme circumstances, surgery to cut the nerve may be needed. A novel approach to target this nervous system using a transcutaneous electrical nerve stimulator (TENS) machine has successfully treated arrhythmias that come from the top chambers of the heart (atrial fibrillation). An ear clip is applied for an hour per day connected to a device (smaller than a phone) that can activate the parasympathetic nervous system (that counteracts the sympathetic nervous system). This is called Low-Level Tragus Stimulation (LLTS). Because it has been used for epilepsy for decades, we have evidence of a very high safety profile and tolerability. We plan to enrol 72 patients, 34 with many PVCs and 38 with VT, and randomise them to either first receive LLTS or first receive sham treatment (this will appear the same to the patient and researchers but without any meaningful vibrations being emitted in the sham group). Each patient will then swap over to the other treatment. We will compare whether the LLTS reduces the amount of ventricular arrhythmias during compared to the amount during the sham treatment period. We will use Holter monitors to measure the amount of PVCs after each period in the PVC group. VT patients have an implantable defibrillator that continuously monitors for VT episodes in this group. We will only enrol adults who can give informed consent, and study participation will not interfere with a patient's clinical treatment.

ELIGIBILITY:
PVC Cohort

Inclusion Criteria:

* Age > 18 years old.
* Participants must understand and be willing to sign a written informed consent document.
* PVC burden of >10% in a 24-hour period on Holter monitoring.

Exclusion Criteria:

* Coronary artery disease
* Known cardiac disease (heart failure or cardiomyopathy) in the documented absence of PVCs. Individuals with suspected PVC-induced cardiomyopathy heart failure, defined as cardiomyopathy or heart failure only diagnosed in the setting of a >10% PVC burden, will be allowed to participate.
* A known diagnosis of Epilepsy.
* Ongoing pregnancy or intention to become pregnant in the forthcoming 12 months.
* Participants using a TENS device for any indication

VT cohort

Inclusion Criteria:

* Participants with structural heart disease and a transvenous implantable cardioverter defibrillator (ICD) in situ
* At least three clinically significant VT events (VT events defined as either >30 seconds of sustained VT, appropriate ICD ATP therapies or appropriate ICD shocks) in the six months before enrolment

Exclusion Criteria:

* Heart failure syndrome with inotrope dependency or requiring mechanical assistance.
* Reversible cause of arrhythmia (e.g. culprit electrolyte abnormality or toxin)
* NYHA (New York Heart Association) stage IV heart failure
* Myocardial infarction or cardiac surgery in the last six months
* Life expectancy <12 months
* Ongoing pregnancy or intention to become pregnant in the forthcoming 12 months.
* Participants using a TENS device for any indication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
VT burden | Six months
  Change in per-subject VT burden as adjudicated by continuous ICD monitoring during the active period versus the sham period (VT burden = the number of ATP events, ICD shocks and sustained (>30 seconds) VT episodes) in the VT cohort
PVC Burden | 14 days
  Change in per-subject PVC burden compared to baseline during the active period versus sham period on 14-day Holter monitoring at the end of the period in the PVC cohort

SECONDARY OUTCOMES:
50% reduction in VT burden | Six months
  The proportion of patients with a 50% reduction in VT burden following LLTS as adjudicated by continuous ICD monitoring (VT burden = number of ATP and ICD shocks and sustained (>30 seconds) VT) in the VT cohort
Change in Kansas City Cardiomyopathy Questionnaire-12 (KCCQ-12) Score in the Active Phase versus Sham Control Phase (VT Cohort) | Six months
  The Kansas City Cardiomyopathy Questionnaire-12 (KCCQ-12) is a validated disease-specific instrument for patients with heart failure. Scores range from 0 to 100, where higher scores indicate better health status, including better symptom control, functional status, and quality of life.
Change in 36-Item Short Form Survey (SF-36) Score in the Active Phase versus Sham Control Phase (PVC Cohort) | 28 days
  The 36-Item Short Form Survey (SF-36) assesses general health-related quality of life. Each domain score and the overall score range from 0 to 100, with higher scores indicating better perceived health and functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Pier D Lambiase, BM BCh, PhD, Principal Investigator — University College, London
Locations (1):
- St Bartholomew's Hospital, Barts Health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No